CLINICAL TRIAL: NCT03093883
Title: Open-label, Randomized, Crossover-design Bioequivalence Study With Comparing a Single Dose of Ferrinemia® Injection With a Single Dose of Venofer® Injection of Vifor AG in Healthy Male Volunteers
Brief Title: Bioequivalence Study Comparing Single Dose of Ferrinemia® Injection With a Single Dose of Venofer® Injection in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azad Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AZAD-BE03; 2016-003602-14 (EudraCT Number)
Record Dates: First submitted 2017-02-16; First posted 2017-03-28 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-07

CONDITIONS: Heathy Volunteers
MeSH Terms: interventions — Ferric Oxide, Saccharated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test product (Experimental): Iron sucrose injection solution 100mg (5 mL single dose vial 20mg/mL elemental iron as iron sucrose for injection).
  Interventions: Drug: Ferrinemia
- Reference product (Active Comparator): Iron sucrose injection solution 100mg (5 mL single dose ampoule 20mg/mL elemental iron as iron sucrose for injection).
  Interventions: Drug: Venofer

INTERVENTIONS:
Drug: Ferrinemia — Test product Ferrinemia will be administered intravenously via a 18 gauge (18G) needle. For intravenous injection, a 5 mL single dose of test product (each mL containing 20 mg/mL elemental iron as iron sucrose in water for injection) will be diluted in 0.9% isotonic sterile sodium chloride (NaCl) up to 15 mL. The injection solution will be intravenously administered to the forearm vein, resulting in a total injection volume of 15 mL administered over a period of 5 minutes.
  Arms: Test product
Drug: Venofer — Reference product Venofer will be administered intravenously via a 18 gauge (18G) needle. For intravenous injection, a 5 mL single dose of test product (each mL containing 20 mg/mL elemental iron as iron sucrose in water for injection) will be diluted in 0.9% isotonic sterile sodium chloride (NaCl) up to 15 mL. The injection solution will be intravenously administered to the forearm vein, resulting in a total injection volume of 15 mL administered over a period of 5 minutes.
  Arms: Reference product

SUMMARY:
The aim of this pharmacokinetic study is to assess the bioequivalence of the generic Ferrinemia® Iron Sucrose injection solution 20 mg/mL manufactured by Help S.A., Greece (test product), to Venofer® Iron Sucrose injection solution 20 mg/mL manufactured by Vifor AG, Switzerland (reference product). Both formulations contain iron as an active ingredient. Intravenous iron sucrose is primarily indicated for the treatment of iron deficiency anemia in adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy volunteers within the age range of 18 to 45 years (both inclusive)
* Comprehension of the nature and purpose of the study and willingness to comply with the requirements of the entire procedure
* Subjects of good health based on previous medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests assessed at the time of screening
* Ferritin levels ≥ 30 µg/l
* Transferrin ≥ 200 mg/dl
* Hemoglobin levels ≥ 13.5 g/dl

Exclusion Criteria:

* Subjects with a BMI of < 19 kg/m2 and > 30 kg/m2
* History of iron deficiency within six months prior screening
* History of anemia within 1 year prior screening
* Presence of iron overload or disturbances in utilization of iron
* History or evidence of allergy or hypersensitivity to the active substance Iron Sucrose of both test and reference product, the finished test and reference product or any of its excipients (water for injection, sodium hydroxide)
* Hypersensitivity to other parenteral iron products
* Use of iron supplements or iron containing herbal or nutritional supplements within last three months prior to start of the study
* History of difficulty with donating blood or difficulty in accessibility of veins in left and right arm
* Donation of blood (one unit or 350 mL) within last three months prior first dose administration of the study drug
* Evidence of an active or suspected cancer, or a history of malignancy within the last 2 years, with the exception of patients with basal cell carcinoma that has been excised and cured
* History of any systemic anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) 6 months prior to the first dose of study drug or the expectation that such treatment will be needed at any time during the study
* History of bleeding disorders or anticoagulant use
* History or other evidence of chronic pulmonary or cardiovascular disease associated with functional limitation
* History of uncontrolled severe seizure disorder
* Any signs of acute infection or inflammation
* History or other evidence of severe illness, or any other condition which would make the subject in the opinion of the investigator, unsuitable for the study.
* Any clinically significant abnormal laboratory values on the laboratory evaluations, medical history or physical examination at the screening
* Positive HIV/HBV/HCV serology tests at the time of the screening visit
* Abnormal 12-lead ECG at the time of screening that is considered to be clinically significant
* History or presence of severe or medical treated allergies or immune or inflammatory conditions (eg. systemic lupus erythematosus, rheumatoid arthritis)
* History of atopic allergy associated with severe asthma
* Recent history or ongoing kidney or liver dysfunction
* Any other major illness in last three months or any significant ongoing chronic medical illness
* Subjects who regularly use more than 2 units of alcohol per day (one unit of alcohol equals ½ liter of beer, 200 mL wine or 50 mL of spirits) or there is evidence of Cocaine, Amphetamines, Methformin, THC, Methadone, MDMA, Morphine, Barbiturates, Benzodiazepines and Tricyclic antidepressants in urine at the screening)
* Heavy smokers (> 10 cigarettes/day) in the last three months prior to start of the study
* Any concomitant medication (except paracetamol) within the last two weeks, including over-the-counter and herbal products, prior to receiving the dose of study medication
* Participation in any clinical trial within last one months
* Subjects who are considered by the investigator to be non-compliant or unlikely to complete the study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Comparative assessment of peak plasma concentration (Cmax) of baseline corrected total serum iron and serum transferrin-bound iron after administration of test and reference product. | -pre-dose -15 minutes and within 5 minutes prior to dosing, at 2, 5, 10, 15, 20, 30, 45 minutes and at 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00, 30.00 hours post-dose.
  bioequivalence between test und reference product of iron sucrose for Cmax of baseline corrected total serum iron and serum transferrin-bound iron.
Comparative assessment of the area under the plasma concentration versus time curve (AUC) of baseline corrected total serum iron and serum transferrin-bound iron after administration of test and reference product. | -pre-dose -15 minutes and within 5 minutes prior to dosing, at 2, 5, 10, 15, 20, 30, 45 minutes and at 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00, 30.00 hours post-dose.
  bioequivalence between test und reference product of iron sucrose for AUC of baseline corrected total serum iron and serum transferrin-bound iron.

SECONDARY OUTCOMES:
Comparative assessment of peak plasma concentration (Cmax) of non-baseline corrected total serum iron and serum transferrin-bound iron after administration of test and reference product. | -pre-dose -15 minutes and within 5 minutes prior to dosing, at 2, 5, 10, 15, 20, 30, 45 minutes and at 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00, 30.00 hours post-dose.
  bioequivalence between test und reference product of iron sucrose for Cmax of non-baseline corrected total serum iron and serum transferrin-bound iron.
Comparative assessment of the area under the plasma concentration versus time curve (AUC) of non-baseline corrected total serum iron and serum transferrin-bound iron after administration of test and reference product. | -pre-dose -15 minutes and within 5 minutes prior to dosing, at 2, 5, 10, 15, 20, 30, 45 minutes and at 1.00, 1.50, 2.00, 3.00, 4.00, 6.00, 8.00, 10.00, 12.00, 24.00, 30.00 hours post-dose.
  bioequivalence between test und reference product of iron sucrose for AUC of non-baseline corrected total serum iron and serum transferrin-bound iron.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No